CLINICAL TRIAL: NCT05473442
Title: A Randomized Phase 2 Study of Adjunctive EQU-001 for Uncontrolled Focal Onset Seizures
Brief Title: Study of EQU-001 for Uncontrolled Focal Onset Seizures
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: insufficient funding to complete the study
Sponsor: Equilibre Biopharmaceuticals B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EQU-202
Record Dates: First submitted 2022-07-18; First posted 2022-07-26 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Focal Onset Seizures
Keywords: EQU-001; Epilepsy; Seizures; Focal; Phase II
MeSH Terms: conditions — Seizures; Epilepsy

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, randomized at a 1:1:1 ratio to receive 20 mg of EQU-001, 60 mg of EQU-001 or a matched placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EQU-001 60 mg (Experimental): EQU-001 60 mg (3 x 20 mg pills)
  Interventions: Drug: EQU-001
- EQU-001 20 mg (Experimental): EQU-001 20 mg (1 x 20 mg pill + 2 x matching placebo pills)
  Interventions: Drug: EQU-001; Other: Matching Placebo
- EQU-001 0 mg (Placebo Comparator): EQU-001 0 mg (3 x matching placebo pills)
  Interventions: Other: Matching Placebo

INTERVENTIONS:
Drug: EQU-001 — 20 mg pills of EQU-001
  Arms: EQU-001 20 mg; EQU-001 60 mg
Other: Matching Placebo — 20 mg matching placebo pills
  Arms: EQU-001 0 mg; EQU-001 20 mg

SUMMARY:
This study is a Phase 2 multinational, double-blind, placebo-controlled, randomized (1:1:1), efficacy and safety study of adjunctive EQU-001 for the treatment of focal onset seizures in subjects aged 18 to 65 years, who have been diagnosed with epilepsy according to International League Against Epilepsy (ILAE) Classification of the Epilepsies 2017 criteria This study is designed to test the efficacy and safety of EQU-001 20 mg and 60 mg as compared with placebo as an add-on anti-seizure medication (ASM) in subjects with uncontrolled focal onset seizures.

The treatment portion of the study will be comprised of a 4-week double-blind medication activation period and a 12-week double-blind maintenance period.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18- 65 years at time of informed consent
2. The subject or designee is willing and able to keep an accurate study diary, the subject is able to adhere to the protocol, the subject or the subject's legal representative is able read, understand, and sign informed consent, as applicable.
3. Diagnosed with focal epilepsy according to ILAE (2017) criteria. Diagnosis to include clinical history and an EEG consistent with focal epilepsy. A normal interictal EEG is allowed when the clinical history is consistent with focal epilepsy.
4. Subject has no seizures that are not focal by the ILAE 2017 criteria
5. Subject must have 8 countable, observable focal seizures during the 8-week baseline period prior to randomization, including at least 3 in each 4-week period with no 21-day seizure-free period. These seizures must be observable (focal aware with motor component, focal impaired awareness, focal to bilateral tonic-clonic) and as such may not include focal aware seizures without a detectable motor component, aphasia, or other observable symptom.
6. Must have had a brain MRI or contrast-enhanced head CT scan with an available report (images need not be available) that has been performed within the past 10 years and that is negative for confounding conditions such as tumor, infection, demyelinating disease, or other progressive neurological disease. Remote stroke that may represent the etiology for epilepsy is allowed. If no such CT or MRI report is available, a potential subject will be asked to undergo a head CT scan with intravenous contrast to meet eligibility criteria prior to study enrollment.
7. Seizures uncontrolled after an adequate trial of at least 1 ASM within the last 2 years.
8. Currently receiving treatment with 1-3 ASMs with doses stable for at least 4 weeks prior to screening. These medications must stay stable during the 8-week baseline period and during the 16-week treatment period. In the case that the plasma level of a concomitant ASM changes, the subject and their physician may then modify the dose to maintain the plasma level that was present prior to beginning the study drug. and must document the change in the EDC system.
9. If participant has a vagal nerve stimulator (VNS), responsive neurostimulator (RNS) or deep brain stimulator (DBS), it must have been implanted and activated >1 year prior to screening, and stimulation parameters that have been stable for >3 months, and battery life of unit anticipated to extend for duration of trial.
10. Females of childbearing potential who are not sexually inactive (abstinent) for 30 days prior to the first dose, throughout the study, and then for 30 days following the last dose, must agree to use of one of the following acceptable birth control methods from 30 days prior to the first dose through 30 days after the last dose of study drug:

    i. Combined estrogen and progestogen containing hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal) together with a condom or other barrier method ii. Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable) together with a condom or other barrier method iii. Intrauterine device (IUD) together with a condom or other barrier method iv. Intrauterine hormone releasing system (IUS) together with a condom or other barrier method v. Bilateral tubal occlusion, hysterectomy, bilateral oophorectomy vi. Vasectomized partner (vasectomy >6 months ago)

For this study, pre-menopausal is defined as not meeting the clinical criteria for post menopausal, that is, no menstrual period for at least one year, in the absence of other identifiable cause(s) of not having a period, together with the absence of typical symptoms of menopause, such as hot flashes and mood instability. True abstinence is allowable when in line with the preferred and usual lifestyle of the subject. Periodic abstinence (such as calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

1. Pregnant or lactating
2. History of hypersensitivity to ivermectin or to any of the excipients in the EQU-001 gelcap
3. History of status epilepticus in the past 1 year from screening
4. History of pseudo- or nonepileptic seizures, or other nonepileptic events that could be confused with epileptic seizures, within the past 5 years
5. History of traumatic brain injury within 30 days prior to screening
6. Resective epilepsy surgery within 1 year; epilepsy-related radiosurgery within 2 years or Ventriculoperitoneal shunt placement within 1 year
7. Presence of progressive neurological disorder or other progressive disorder or unstable medical condition(s) that may confound study results. History of long QT syndrome, family history of sudden death of unknown cause.
8. Psychiatric disorder where changes in pharmacotherapy are needed or anticipated during the study or which would interfere with the subject's ability to participate in the trial
9. Active suicidal plan/intent in the past 6 months, a history of suicide attempt in the last 2 years, or more than 1 lifetime suicide attempt as evidenced by a positive response to C-SSRS questions 4 or 5
10. History of substance use disorder, including alcohol, within the past 2 years
11. Currently in another investigational drug study
12. Currently on felbamate for less than one year before visit 1 (aplastic anemia and hepatic failure usually occur within 6 months to one year). If on felbamate, documentation of stable hemogram and liver enzyme tests must be present.
13. Currently on vigabatrin for less than 2 years before visit 1, as most visual field changes occur between 6 months and 2 years Subjects on vigabatrin should have available, appropriate documentation of visual fields.
14. Currently taking retigabine/ezogabine
15. History of intermittent use of rescue benzodiazepines (i.e., 1 to 2 doses over a 24-hour period is considered a 1-time rescue) more than once in the 4 weeks prior to the baseline visit or more than once per 4 weeks during the 8-week baseline period If a subject is taking benzodiazepines for an indication other than epilepsy (e.g., anxiety, sleep), the dose should to be stable for at least 4 weeks prior to screening and remain stable throughout screening and double blind periods of the study.
16. Currently taking ivermectin, or has taken it within the last 4 weeks prior to visit 1

17a. Use of the following medications within 4 weeks of the baseline visit and throughout the study that may interfere with study drug metabolism (please note ASMs with CYP3A4 metabolism are not excluded from this study, as drug levels and safety are monitored throughout the study):

i. CYP3A4 inducers: rifampin, lumacaftor, mitotane, enzalutamide, apalutamide, St. John's wort, glucocorticoids

ii. Medications with PGP interactions: amiodarone, apalutamide, verapamil, lorlatinib, rifampin, St. John's wort

17b. Use of the following medications/foods is not strictly prohibited but is discouraged. Please make every attempt to refrain and to record each incidence of use of any of these (along with all medications and supplements):

i. CYP3A4 inhibitors, including, but not limited to clarithromycin, ceritinib, idelalisib, lonafarnib, tucatinib, erythromycin, telithromycin, diltiazem, dronedarone, posaconazole, voriconazole, nefazodone, itraconazole, ketoconazole, anti-retroviral drugs (atazanavir, darunavir, indinavir, lopinavir, nelfinavir, ritonavir, saquinavir, tipranavir), grapefruit and grapefruit juice, pomegranate fruit and pomegranate juice

ii. Additional medications that may interact with CYP3A4, PGP, or Vitamin K: fluconazole, isavuconazole, cyclosporine, dronedarone, imatinib, warfarin, acenocoumarol

18. Has any of the following laboratory or exam abnormalities: i. Positive urine drug screen (methamphetamines, amphetamines, cocaine, PCP, opioids, barbiturates) at screening without a therapy related explanation ii. Positive hCG (female participants) (at screening or visit 2/enrollment) iii. QTcF > 450 msec at visit 2/enrollment

19. Subject is not approved for study inclusion by the Epilepsy Consortium based on the diagnostic review form

20. Any condition that, in the opinion of the investigator, may impact a subject's safety or ability to follow study procedures

21. History of 14 or more consecutive days in Angola, Equatorial Guinea, Gabon, Cameroon, the Central African Republic, the Republic of Congo, the DR of Congo, Nigeria, Chad, and/or South Sudan within the past 17 years and did not take diethylcarbamazine prophylaxis or has not been evaluated for/found to be negative for or treated for loa loa and subsequently evaluated as resolved since the most recent stay of at least 14 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-12-27 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Median percentage change in the overall number of countable observable seizures | Every 4 weeks from week 1 up to week 16
  per 28-day period relative to baseline in each treatment arm during the double-blind treatment period compared with placebo.

SECONDARY OUTCOMES:
Median percentage change in the overall number of countable observable seizures | Every 4 weeks from week 5 up to week 16
  per 28-day period relative to baseline in each treatment arm during the maintenance phase compared with placebo
≥ 50% responder rates | Week 1 to 16
  In the treated arms as compared with placebo during double blind components of the study, which consist of the medication activation and maintenance period
≥ 50% responder rates | Week 5 to 16
  In the treated arms as compared with placebo during the maintenance period alone
Difference in PGI-C Scale: Patient's Global Impression of Change (PGIC) | Week 6 to 16
  In each treated cohort as compared with placebo at days 42 and 112. PGI-C Scale ranges from 'Very much improved' to 'Very much worse'
Median percentage change in the number of countable observable seizures by subtype | Week 1 to 16
  Subtype (focal aware with motor component, focal impaired aware, and focal to bilateral tonic-clonic) per 28 days during the maintenance period (treatment weeks 5-16) and during the entire double blind period in the treated and placebo arms
Percent (%) of subjects who are seizure free | Week 5 to 16
  by study days 29-112
Percent (%) of subjects who are seizure free in treated arms as compared with placebo | Week 5 to 16
≥ 70% and ≥ 90% response rates in treated arms compared with placebo | Week 5 to 16
  during the maintenance period
Change from visit 2 (enrollment) in the Patient weighted Quality of Life in Epilepsy (QOLIE 31-P) scale score | Week 6 to 16
  at days 42 and 112 in each treated arm as compared with placebo
Number of subjects who withdraw from treatment | Week 1 to 16
  because of an AE in each treatment arm
Number of adverse events (CTCAE grade 2 or higher) | Week 1 to 16
  in the treatment arms compared with placebo
Change in Columbia-Suicide Severity Rating Scale (C-SSRS) | Week 1 to 16
  from visit 2 in each treated arm as compared with placebo at each measured timepoint

CONTACTS AND LOCATIONS:
Locations (13):
- United States (8):
  - Consultants in Epilepsy and Neurology, PLLC, Boise, Idaho
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Institute of Neurology and Neurosurgery at Saint Barnabas, Livingston, New Jersey
  - NYU Langone Health, New York, New York
  - Sooner Clinical Research, Inc., Oklahoma City, Oklahoma
  - Comprehensive Epilepsy Center at Thomas Jefferson University, Philadelphia, Pennsylvania
  - Northwest Houston Neurology, Cypress, Texas
  - University of Virginia, Charlottesville, Virginia
- Israel (5):
  - Ramban Health Care Campus, Haifa
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv